CLINICAL TRIAL: NCT06336070
Title: Postmenopausal Oncological Women Exercising for Recover Their Health. Associations and Changes in Metabolic Flexibility and Autonomic Control After Two Training Programs (Muscle Power vs Metabolic Power): the POWER Health Study
Brief Title: Metabolic Flexibility and Autonomic Control After Muscle Power vs Metabolic Power Training in Postmenopausal Oncological Women: the POWER Health Study
Acronym: POWER Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Generalitat Valenciana (Other)
Responsible Party: Principal Investigator, Cristina Blasco-Lafarga, Senior Lecturer, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-FIS-3251696; CIACIF/2022/368 (Other Grant/Funding Number: Regional Ministry of Education, Universities and Employment - Generalitat Valenciana)
Record Dates: First submitted 2024-03-14; First posted 2024-03-28 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer Female; Cardiometabolic Syndrome; Metabolism Disorder, Lipid; Autonomic Dysfunction; Cardiovascular Diseases in Old Age
Keywords: Metabolic Flexibility; Heart Rate Variability; Muscle Power; Resting metabolic Rate; Lactate; High Intensity Interval Training; Strength Training; Breast Cancer; Ageing; Menopause; Female; Exercise Training
MeSH Terms: conditions — Metabolic Syndrome; Lipid Metabolism Disorders; Primary Dysautonomias; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Two cohorts of both healthy postmenopausal women and women free of postmenopausal breast cancer recurrence. Each of the groups will be split into two different exercise programmes. Both programmes, High Intensity Interval Training (HIIT) programme (metabolic power training) and Muscle Power Intervention (MPI) programme will consist of 8 weeks.
  Interventions: Behavioral: HIIT program (8 weeks); Behavioral: MPI program (8 weeks)
- Control group (No Intervention): Two cohorts of both healthy postmenopausal women and women free of postmenopausal breast cancer recurrence.

INTERVENTIONS:
Behavioral: HIIT program (8 weeks) — Metabolic Power Training: A High Intensity Interval Training (HIIT) intervention, 3 times per week (30 min session) during 8 weeks with professional supervision and intensities adapted and modified during the intervention period.
  Arms: Exercise group
Behavioral: MPI program (8 weeks) — Muscle Power Intervention (MPI), 2 times per week (45 min session) during 8 weeks with professional supervision and intensities adapted and modified during the intervention period.
  Arms: Exercise group

SUMMARY:
POWER Health is a randomized clinical trial with a two-arm parallel design whose objectives are 1) to study metabolic flexibility and autonomic function (both capacities that describe cardiovascular health) in a sample of postmenopausal oncological women vs postmenopausal untreated controls (CT); and 2) to analyze the impact of two different 8-week physical exercise supervised interventions: HIIT training vs strength training focused on muscle power, on both cardiovascular capacities in these populations.

DETAILED DESCRIPTION:
Nowadays, breast cancer is the most common type of cancer worldwide, accounting for 30% of all cancers in Spanish women in 2023. Cancer is also the second leading cause of death in developed countries, following cardiovascular diseases, with which it shares a close relationship. Additionally, we know that the incidence of breast cancer increases with age, experiencing a rise after menopause. However, lifestyle and physical exercise are known to improve the prevention, prognosis, and survival of this disease, as well as enhance quality of life in these patients. Indeed, recent studies have highlighted the relevance of cardiovascular health in this oncological process, as well as the potential of physical exercise interventions to improve cardiovascular health following the disease.

POWER Health is a randomized clinical trial aimed at studying metabolic flexibility and autonomic health in a population of breast cancer recurrence-free women (RFC) compared to postmenopausal untreated controls (CT), along with the implementation of two supervised exercise interventions in both populations. These interventions will last for 8 weeks, one involving HIIT exercise focused on improving metabolic power (MPI), and the other one involving strength exercise focused on enhancing muscular power, with the hypothesis of better metabolic flexibility and autonomic function, and consequently, better cardiovascular health.

POWER health is a mixed method design: cross-sectional & longitudinal study. Given the feasibility and simple application of POWER Health, this clinical trial will contribute to the prevention and improvement of the health of postmenopausal women, with an important clinical and economic impact, not only in the scientific community but also in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed of relapse free-cancer (RFC) or patients not diagnosed of any cancer at least the last 15 years (CG)
* Aged between 35 and 75 years
* Diagnostic of breast cancer (i.e., including ductal carcinoma, invasive carcinoma, triple negative; RFC) or physiological menopause (CG)
* Not participating in a nutritional/dietary intervention
* Not being physically active (i.e., not to be participating in any physical exercise program in the last 3 months, or performing less than 600 metabolic equivalents (METS)/week of moderate-vigorous physical activity).
* To be capable and willing to provide informed consent
* Not to suffer from any specific condition that may impede testing of the study hypothesis or make it unsafe to engage in the exercise intervention (i.e., determined by the research staff).

Exclusion Criteria:

* Medical contraindication for being engaged in an exercise.
* Additional surgery planned within the intervention
* Consuming usually betablocker or any drugs alterning nervous system functioning
* History of another primary invasive cancer (RFC) or suffer a serious chronic illness (CG)
* To present any of the following cardiac conditions: (i) myocardial infarction or coronary revascularization procedure within prior 3 months, (ii) uncontrolled hypertension (i.e., systolic ≥180 mmHg or diastolic ≥100 mmHg), (iii) uncontrolled arrhythmias (iv) valvular disease clinically significant, (v) decompensated heart failure or (vi) to suffer from known aortic aneurysm.

Ages: 35 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Fat oxidation during incremental test | Preintervention (only this one in cross-sectional study) and Postintervention (8 weeks after)
  Fat oxidation rates calculated from VO2 and VCO2 values collected by indirect calorimetry (COSMED K5 portable metabolic analyzer, Rome, Italy) and after applying Frayn's stoichiometric formulae, during an incremental test from 0.45 W/kg with 0.15W/kg each 4-min step
Detrended Fluctuation Analysis | Preintervention and Postintervention (8 weeks after)
  Non-linear mathematical variable that allows collecting physiological information and vagal activity of the organism, analysed in 2-minute intervals by Kubios Scientific software (Kuopio, Finland), during the incremental test

SECONDARY OUTCOMES:
Weight | Preintervention and Postintervention (8 weeks after)
  Weight measured with a scale (kg)
Height | Preintervention and Postintervention (8 weeks after)
  Height measured with a stadiometer (cm)
Calf, waist and hip circumferences. | Preintervention and Postintervention (8 weeks after)
  Calf, waist and hip circumferences will be assessed with an anthropometric tape measure (cm)
Lean mass | Preintervention and Postintervention (8 weeks after)
  Body composition assessment will be obtained by bioimpedance (Tanita DC-430 MA S; Tokyo, Japan; kg)
Fat-free mass | Preintervention and Postintervention (8 weeks after)
  Body composition assessment will be obtained by bioimpedance (Tanita DC-430 MA S; Tokyo, Japan; kg)
Visceral adipose tissue | Preintervention and Postintervention (8 weeks after)
  Body composition assessment will be obtained by bioimpedance (Tanita DC-430 MA S; Tokyo, Japan; kg)
Bone Mass | Preintervention and Postintervention (8 weeks after)
  Body composition assessment will be obtained by bioimpedance (Tanita DC-430 MA S; Tokyo, Japan; kg)
Fat mass | Preintervention and Postintervention (8 weeks after)
  Body composition assessment will be obtained by bioimpedance (Tanita DC-430 MA S; Tokyo, Japan; kg)
Blood Pressure | Preintervention and Postintervention (8 weeks after)
  The investigators will also assess systolic and diastolic blood pressure in the left (whenever possible) arm at rest.
Oxygen Saturation | Preintervention and Postintervention (8 weeks after)
  The investigators will also assess oxygen saturation in middle finger of the right hand at rest.
Sarcopenia | Preintervention and Postintervention (8 weeks after)
  The SARC-F will be used to evaluate the risk of sarcopenia
Physical activity and sedentariness | Preintervention and Postintervention (8 weeks after)
  The International Physical Activity Questionnaire (IPAQ) will be used to evaluate the current physical activity level of the participants. Minimum value = 0 min/day of physical activity // Maximum value = 1440 min/day of physical activity. Higher scores imply a more physically active pattern.
Lactate | Preintervention and Postintervention (8 weeks after)
  Lactate assessment will be obtained by lactate analyzer (Lactate Scout Sport SensLab GmbH, Leipzig, Germany)
Rating Perceived Exertion | Preintervention and Postintervention (8 weeks after)
  The Rating Perceived Exertion (RPE) of Borg scale will be used to obtain the perceived effort. Minimum value: 1 // Maximum value: 10. Higher scores mean a worse outcome.
Visual Analogue Scale of Pain | Preintervention and Postintervention (8 weeks after)
  The Visual Analogue Scale of Pain (VAS) scale will be used to obtain the local pain assessment. Minimum value: 1 // Maximum value: 10. Higher scores mean a worse outcome.
Cadence | Preintervention and Postintervention (8 weeks after)
  Cadence will be monitorized by the smart roller Saris H3 (CycleOps Hammer Direct Drive Trainer, Saris, Madison, USA).
Mechanical Power | Preintervention and Postintervention (8 weeks after)
  Power will be monitorized by the smart roller Saris H3 (CycleOps Hammer Direct Drive Trainer, Saris, Madison, USA).
Muscle Power 5STS | Preintervention and Postintervention (8 weeks after)
  Power will be calculated by Power Frail App (Toledo, Spain)
Basal metabolic rate | Preintervention and Postintervention (8 weeks after)
  Metabolic rate will be registered by indirect calorimetry (COSMED K5 portable metabolic analyzer, Rome, Italy) in baseline conditions
Respiratory exheange ratio at rest | Preintervention and Postintervention (8 weeks after)
  Resting exchange ratio will be registered by indirect calorimetry (COSMED K5 portable metabolic analyzer, Rome, Italy) in baseline conditions
Fat oxidation at rest | Preintervention and Postintervention (8 weeks after)
  Fat oxidation will be registered by indirect calorimetry (COSMED K5 portable metabolic analyzer, Rome, Italy) in baseline conditions
Carbohydrate oxidation at rest | Preintervention and Postintervention (8 weeks after)
  Carbohydrate will be registered by indirect calorimetry (COSMED K5 portable metabolic analyzer, Rome, Italy) in baseline conditions
Carbohydrate oxidation during incremental test | Preintervention and Postintervention (8 weeks after)
  Carbohydrate oxidation rates will be calculated from VO2 and VCO2 values collected by indirect calorimetry (COSMED K5 portable metabolic analyzer, Rome, Italy) and after applying Frayn's stoichiometric formulae, during an incremental test from 0.45 W/kg with 0.15W/kg each 4-min step
Energy expenditure during incremental test | Preintervention and Postintervention (8 weeks after)
  Energy expenditure rate will be calculated will be collected by indirect calorimetry (COSMED K5 portable metabolic analyzer, Rome, Italy) during an incremental test
FATmax intensity | Preintervention and Postintervention (8 weeks after)
  FATmax will be calculated will be collected by indirect calorimetry (COSMED K5 portable metabolic analyzer, Rome, Italy) during an incremental test
VO2peak | Preintervention and Postintervention (8 weeks after)
  VO2peak will be calculated will be collected by indirect calorimetry (COSMED K5 portable metabolic analyzer, Rome, Italy) during an incremental test
Sample Entropy | Preintervention and Postintervention (8 weeks after)
  Non-linear mathematical variable that allows collecting physiological information and parasympathetic activity of the organism, analysed in 3-minute intervals by Kubios Scientific software (Kuopio, Finland), during the incremental test
SD1/SD2 ratio | Preintervention and Postintervention (8 weeks after)
  Linear mathematical variable that allows collecting physiological information and parasympathetic activity of the organism, analysed in 2-minute intervals by Kubios Scientific software (Kuopio, Finland), during the incremental test
The root mean square of successive differences between normal heartbeats (RMSSD) | Preintervention and Postintervention (8 weeks after)
  Linear mathematical variable that allows collecting physiological information and parasympathetic activity of the organism, analysed in 2-minute intervals by Kubios Scientific software (Kuopio, Finland), during the incremental test

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Blasco Lafarga, Tenured Professor, Principal Investigator — University of Valencia
Locations (1):
- Faculty of Physical Activity and Sport Sciences, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Monferrer-Marin J, Roldan A, Monteagudo P, Chulvi-Medrano I, Blasco-Lafarga C. Impact of Ageing on Female Metabolic Flexibility: A Cross-Sectional Pilot Study in over-60 Active Women. Sports Med Open. 2022 Jul 30;8(1):97. doi: 10.1186/s40798-022-00487-y. PMID 35907092
- [Result] Blasco-Lafarga C, Monferrer-Marin J, Roldan A, Monteagudo P, Chulvi-Medrano I. Metabolic Flexibility and Mechanical Efficiency in Women Over-60. Front Physiol. 2022 Apr 6;13:869534. doi: 10.3389/fphys.2022.869534. eCollection 2022. PMID 35464093
- [Result] Frandsen J, Amaro-Gahete FJ, Landgrebe A, Dela F, Ruiz JR, Helge JW, Larsen S. The influence of age, sex and cardiorespiratory fitness on maximal fat oxidation rate. Appl Physiol Nutr Metab. 2021 Oct;46(10):1241-1247. doi: 10.1139/apnm-2021-0080. Epub 2021 Apr 13. PMID 33848440
- [Result] Gonzalez-Acedo A, Plaza-Florido A, Amaro-Gahete FJ, Sacha J, Alcantara JMA. Associations between heart rate variability and maximal fat oxidation in two different cohorts of healthy sedentary adults. Nutr Metab Cardiovasc Dis. 2022 Oct;32(10):2338-2347. doi: 10.1016/j.numecd.2022.06.015. Epub 2022 Jun 22. PMID 35977864
- [Result] Smith RL, Soeters MR, Wust RCI, Houtkooper RH. Metabolic Flexibility as an Adaptation to Energy Resources and Requirements in Health and Disease. Endocr Rev. 2018 Aug 1;39(4):489-517. doi: 10.1210/er.2017-00211. PMID 29697773
- [Result] Sogaard D, Lund MT, Scheuer CM, Dehlbaek MS, Dideriksen SG, Abildskov CV, Christensen KK, Dohlmann TL, Larsen S, Vigelso AH, Dela F, Helge JW. High-intensity interval training improves insulin sensitivity in older individuals. Acta Physiol (Oxf). 2018 Apr;222(4):e13009. doi: 10.1111/apha.13009. Epub 2017 Dec 19. PMID 29197155
- [Result] Formighieri C, Muller DC, Saez de Asteasu ML, Mello A, Teodoro JL, Boeno F, Grazioli R, Cunha GDS, Pietta-Dias C, Izquierdo M, Pinto RS, Cadore EL. Interindividual variability of adaptations following either traditional strength or power training combined to endurance training in older men: A secondary analysis of a randomized clinical trial. Exp Gerontol. 2022 Nov;169:111984. doi: 10.1016/j.exger.2022.111984. Epub 2022 Oct 19. PMID 36270544
- [Result] Mugele H, Freitag N, Wilhelmi J, Yang Y, Cheng S, Bloch W, Schumann M. High-intensity interval training in the therapy and aftercare of cancer patients: a systematic review with meta-analysis. J Cancer Surviv. 2019 Apr;13(2):205-223. doi: 10.1007/s11764-019-00743-3. Epub 2019 Feb 26. PMID 30806875
- [Result] Toohey K, Pumpa K, McKune A, Cooke J, Welvaert M, Northey J, Quinlan C, Semple S. The impact of high-intensity interval training exercise on breast cancer survivors: a pilot study to explore fitness, cardiac regulation and biomarkers of the stress systems. BMC Cancer. 2020 Aug 20;20(1):787. doi: 10.1186/s12885-020-07295-1. PMID 32819304
- [Result] Matsubara Y, Kiyohara H, Teratani T, Mikami Y, Kanai T. Organ and brain crosstalk: The liver-brain axis in gastrointestinal, liver, and pancreatic diseases. Neuropharmacology. 2022 Mar 1;205:108915. doi: 10.1016/j.neuropharm.2021.108915. Epub 2021 Dec 15. PMID 34919906